CLINICAL TRIAL: NCT02428855
Title: Phase II Trial of Dasatinib in Patients With Isocitrate Dehydrogenase (IDH)-Mutant Advanced Intrahepatic Cholangiocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry); TargetCancer Foundation (Other)
Responsible Party: Principal Investigator, Bruce Giantonio, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-007
Record Dates: First submitted 2015-04-23; First posted 2015-04-29 (Estimated); Results first posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasatinib (Experimental): Patients with advanced intrahepatic cholangiocarcinoma who have either IDH1 or IDH2 mutations and have received at least one prior platinum containing regimen
  * Dasatinib, oral, daily, predetermined dosage per cycle
  * Radiologic Response Assessment every 2 cycles
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib
  Other Names: SPRYCEL ™

SUMMARY:
This research study is studying Dasatinib as a possible treatment for cancer of bile ducts.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The standard treatment for metastatic cholangiocarcinoma is combination chemotherapy with gemcitabine and cisplatin. The FDA (the U.S. Food and Drug Administration) has not approved dasatinib for your specific disease (Cholangiocarcinoma) but it has been approved for other uses (Chronic Myeloid Leukemia)

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Participants must have unresectable or metastatic histologically confirmed intrahepatic cholangiocarcinoma
* Patients must have either IDH1 or IDH2 mutations (any known mutations) based on the SNaPshot platform or other molecular testing platform from either archived tissue or fresh biopsy (tested in CLIA-certified lab)
* Patients with other biliary tract cancers (extrahepatic or gallbladder cancers) with IDH1 or IDH2 mutations are allowed
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥10 mm with spiral CT scan. See section 10 for the evaluation of measureable disease.
* Participants must have received at least one prior platinum-based regimen for advanced cholangiocarcinoma and had progressive disease or become intolerable to the regimen
* Age ≥18 years.
* Life expectancy of ≥3 months.
* ECOG performance status 0 or 1 (see Appendix A).
* Participants must have adequate organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,200/mcL
  * Platelets ≥75,000/mcL
  * Hemoglobin ≥9 g/dL
  * Total bilirubin ≤ 2.5 x the upper limit of normal
  * AST (SGOT)/ALT (SGPT) ≤ 5 X institutional upper limit of normal
  * PT/PTT ≤ 1.5 x ULN
  * Creatinine ≤ 1.5 or GFR ≥ 60 mL/min/1.73m2
  * Serum Albumin ≥2.8 g/dl
* Prior chemoembolization, radiofrequency ablation, or radiation to the liver is allowed as long as the patient has measurable disease outside of the treated area or measurable progression at the site of the treated area
* Ability to understand and the willingness to sign a written informed consent document.
* Sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (eg, male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s).
* Women of childbearing potential must have a negative pregnancy test at screening. Women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal. Postmenopause is defined as amenorrhea ≥ 12 consecutive months. Note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, ovarian suppression or any other reversible reason.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Prior treatment with dasatinib
* Periampullary tumors
* Chemotherapy, within 4 weeks prior to entering the study (6 weeks for nitrosoureas or mitomycin) or those who have not recovered to less than or equal to grade 1 from adverse events due to agents administered more than 4 weeks earlier.
* The subject has received radiation therapy:

  * to bone or brain metastasis within 14 days of the first dose of study treatment
  * to any other site(s) within 28 days of the first dose of study treatment
* The subject has active brain metastases or epidural disease (Note: Subjects with brain metastases previously treated with whole brain radiation or radiosurgery or subjects with epidural disease previously treated with radiation or surgery who are asymptomatic and do not require steroid treatment for at least 2 weeks before starting study treatment are eligible. Neurosurgical resection of brain metastases or brain biopsy is permitted if completed at least 3 months before starting study treatment. (Baseline brain imaging with contrast-enhanced CT or MRI scans for subjects with known brain metastases is required to confirm eligibility.)
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including

    * Congestive heart failure (CHF): New York Heart Association (NYHA) Class III (moderate) or Class IV (severe) at the time of screening
    * Concurrent uncontrolled hypertension defined as sustained BP > 140 mm Hg systolic, or > 90 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment
    * Diagnosed or suspected congenital long QT syndrome
    * Any of the following within 6 months before the first dose of study treatment:

      * Unstable angina pectoris
      * Clinically-significant cardiac arrhythmias
      * Stroke (including TIA, or other ischemic event)
      * Myocardial infarction
      * Thromboembolic event requiring therapeutic anticoagulation (Note: subjects with a venous filter (e.g. vena cava filter) are not eligible for this study)
      * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes)
      * Prolonged QTc interval on pre-entry electrocardiogram (> 450 msec), may use either the Fridericia and Bazett's correction
      * Hypokalemia or hypomagnesemia that is not corrected prior to dasatinib administration
      * Patients should not be taking drugs that are generally accepted to have a risk of causing Torsades de Pointes. The following must be discontinued at least 7 days prior to starting dasatinib to be eligible:quinidine, procainamide, disopyramide, amiodarone, sotalol, ibutilide,dofetilide, erythromycins, clarithromycin, chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide, cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine,levomethadyl, pentamidine, sparfloxacin, lidoflazine
  * Other clinically significant disorders such as:

    * active infection requiring systemic treatment within 28 days before the first dose of study treatment
    * serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
  * Patients with known moderate/severe pleural effusions that are unrelated to malignancy or established diagnosis of pulmonary arterial hypertension
* Concurrent malignancy (other than adequately treated non-melanoma skin cancer, superficial transitional cell carcinoma of the bladder, and cervical carcinoma in situ) diagnosed within the past 3 years or any currently active malignancy
* Psychiatric illness/social situations that would limit compliance with study requirements.
* The subject has received any other type of investigational agent within 28 days before the first dose of study treatment.
* The subject is unable to swallow tablets
* Individuals who are known to be HIV-positive are excluded from this study.
* Pregnant women are excluded from this study due to the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with dasatinib, breastfeeding should be discontinued if the mother is treated with dasatinib. These potential risks may also apply to other agents used in this study.
* Subjects may not be receiving any other study agents concurrently while on this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Giantonio, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Groups:
- Dasatinib: Patients with advanced intrahepatic cholangiocarcinoma who have either IDH1 or IDH2 mutations and have received at least one prior platinum containing regimen
  * Dasatinib, oral, daily, predetermined dosage per cycle
  * Radiologic Response Assessment every 2 cycles
  Dasatinib
Period: Overall Study
Arm/Group | Dasatinib
Started | 8
Completed | 6
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Dasatinib
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 59 [45 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 8
Tumor location [Count of Participants; unit: Participants]
  Intrahepatic | 7
  Hilar | 1
IDH Mutation [Count of Participants; unit: Participants]
  IDH1 | 7
  IDH2 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: The number of participants that achieved either a complete or partial response, as assessed by Response Criteria in Solid Tumors (RECIST 1.1)
  * Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 8 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 8
Participants
  Complete Response (CR) | 0
  Partial Response (CR) | 0

2. Secondary Outcome: Median Progression Free Survival (PFS)
Description: The median amount of time from registration until disease progression or death, whichever occurs first. Disease progression was assessed via RECIST 1.1 criteria:
  > Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From registration until disease progression or death, median duration of 8.7 weeks
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Dasatinib
Number analyzed (Participants) | 8
Weeks | 8.7 [6.4 to NA] — Upper limit of the confidence interval is not defined due to an insufficient number of events occurring.

3. Secondary Outcome: Overall Survival
Description: The median amount of time from registration until death. Participants are censored at the date last known alive.
Time Frame: From the time of registration until death, median duration of 37.9 weeks
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Dasatinib
Number analyzed (Participants) | 8
Weeks | 37.9 [20.7 to NA] — The upper limit of the confidence interval is not defined due to an insufficient number of events occurring.

4. Secondary Outcome: Number of Participants With Adverse Events
Description: The number of participants that experienced an adverse event as assessed by Common Toxicology Criteria for Adverse Events (CTCAE 4.0)
Time Frame: From the start of treatment until 30 days after the end of treatment, median duration of 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 8
Participants | 8

ADVERSE EVENTS:
Time Frame: From the start of treatment until 30 days after the end of treatment, median duration of 3 months
Description: Only grade 3 or greater treatment related adverse events were recorded
Arm/Group | Dasatinib
All-Cause Mortality (participants affected / at risk) | 7/8
Serious Adverse Events (participants affected / at risk) | 8/8
Other Adverse Events (participants affected / at risk) | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=8)
Lymphopenia (Blood and lymphatic system disorders) | 4
Anemia (Blood and lymphatic system disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Menorrhagia (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT02428855/Prot_SAP_000.pdf